CLINICAL TRIAL: NCT06582056
Title: A Multi-center, Cross-sectional Study to Investigate Immunological, Clinical, and Microbiological Biomarkers in Well-characterized Populations With or Without Periodontitis and/or Type 2 Diabetes Mellitus in Male and Female Participants Aged 30 -70 Years
Brief Title: Study on Biomarkers of Periodontitis and Type 2 Diabetes Mellitus in Males and Females 30 - 70 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VPE00001; U1111-1306-7393 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-07-30; First posted 2024-09-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Periodontal Disease
Keywords: Type 2 diabetes mellitus; Porphyromonas gingivalis
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Healthy Participant or Participant with Gingivitis with no Type 2 Diabetes Mellitus (Other): Participants will be screened via periodontal exam for periodontal disease staging and point-of-care hemoglobin A1c (HbA1c) testing for type 2 diabetes (T2DM) status. Blood, saliva, subgingival plaque, and gingival crevicular fluid (GCF) will be collected
  Interventions: Procedure: Investigational Procedure
- Healthy Participant or Participant with Gingivitis with Hemoglobin A1c level 6.5-7.8 (Other): Participants will be screened via periodontal exam for periodontal disease staging and point-of-care hemoglobin A1c (HbA1c) testing for type 2 diabetes (T2DM) status. Blood, saliva, subgingival plaque, and gingival crevicular fluid (GCF) will be collected
  Interventions: Procedure: Investigational Procedure
- Healthy Participant or Participant with Gingivitis with Hemoglobin A1c level 8.0-10.0 (Other): Participants will be screened via periodontal exam for periodontal disease staging and point-of-care hemoglobin A1c (HbA1c) testing for type 2 diabetes (T2DM) status. Blood, saliva, subgingival plaque, and gingival crevicular fluid (GCF) will be collected
  Interventions: Procedure: Investigational Procedure
- Participant with Stage I/Stage II Periodontal Disease with no Type 2 Diabetes Mellitus (Other): Participants will be screened via periodontal exam for periodontal disease staging and point-of-care hemoglobin A1c (HbA1c) testing for type 2 diabetes (T2DM) status. Blood, saliva, subgingival plaque, and gingival crevicular fluid (GCF) will be collected
  Interventions: Procedure: Investigational Procedure
- Participant with Stage I/Stage II Periodontal Disease with Hemoglobin A1c level 6.5-7.8 (Other): Participants will be screened via periodontal exam for periodontal disease staging and point-of-care hemoglobin A1c (HbA1c) testing for type 2 diabetes (T2DM) status. Blood, saliva, subgingival plaque, and gingival crevicular fluid (GCF) will be collected
  Interventions: Procedure: Investigational Procedure
- Participant with Stage I/Stage II Periodontal Disease with Hemoglobin A1c level 8.0-10.0 (Other): Participants will be screened via periodontal exam for periodontal disease staging and point-of-care hemoglobin A1c (HbA1c) testing for type 2 diabetes (T2DM) status. Blood, saliva, subgingival plaque, and gingival crevicular fluid (GCF) will be collected
  Interventions: Procedure: Investigational Procedure
- Participant with Stage III/Stage IV Periodontal Disease with no Type 2 Diabetes Mellitus (Other): Participants will be screened via periodontal exam for periodontal disease staging and point-of-care hemoglobin A1c (HbA1c) testing for type 2 diabetes (T2DM) status. Blood, saliva, subgingival plaque, and gingival crevicular fluid (GCF) will be collected
  Interventions: Procedure: Investigational Procedure
- Participant with Stage III/Stage IV Periodontal Disease with Hemoglobin A1c level 6.5-7.8 (Other): Participants will be screened via periodontal exam for periodontal disease staging and point-of-care hemoglobin A1c (HbA1c) testing for type 2 diabetes (T2DM) status. Blood, saliva, subgingival plaque, and gingival crevicular fluid (GCF) will be collected
  Interventions: Procedure: Investigational Procedure
- Participant with Stage III/Stage IV Periodontal Disease with Hemoglobin A1c level 8.0-10.0 (Other): Participants will be screened via periodontal exam for periodontal disease staging and point-of-care hemoglobin A1c (HbA1c) testing for type 2 diabetes (T2DM) status. Blood, saliva, subgingival plaque, and gingival crevicular fluid (GCF) will be collected
  Interventions: Procedure: Investigational Procedure

INTERVENTIONS:
Procedure: Investigational Procedure — It consists of prospective blood and/or tissue collection from healthy subjects and/or patients with the appropriate clinical annotation. Study without any IMP administration.

SUMMARY:
The purpose of this study is to learn about the interactions of markers of type 2 diabetes (T2DM) and periodontitis (PD). Study VPE00001 is a multi-center cross-sectional study. Participants will be categorized based on point-of-care hemoglobin A1c (HbA1c) and periodontal disease (PD) staging into 9 subgroups. The key objectives of the study are:

* To evaluate immune signatures in well-characterized populations with or without PD and/or T2DM
* To evaluate baseline clinical biomarkers of T2DM and PD in well-characterized populations
* To evaluate the influence of clinical, immunological, and microbiological biomarkers on the bidirectional relationship between T2DM and PD

DETAILED DESCRIPTION:
The duration of each participant will be up to 30 days with a screening visit and a single visit for specimen collection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 to 70 years on the day of inclusion (30 to 70 years means from the day of the 30th birthday to the day before the 71st birthday)
* Body mass index < 40 kg/m2
* Participants without type 2 diabetes mellitus (T2DM) or pre-diabetes (as confirmed by hemoglobin A1C (HbA1c) < 5.7%) or Participants diagnosed with T2DM for at least 6 months with HbA1c between 6.5%-7.8% or 8%-10% on the day of screening
* Participants without PD (healthy or with gingivitis), or participants diagnosed with stages I/II or stages III/IV PD within 2 weeks of sample collection

Exclusion Criteria:

* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating blood sampling
* History of human immunodeficiency virus (HIV) infection, or active hepatitis B (HB) or hepatitis C virus infection
* Known or recently active (within 12 months) neoplastic disease (including skin cancer) or a current or past diagnosis of any hematologic malignancy (ie, leukemia)
* Participants with pre-existing unstable disease, defined as disease requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks prior to enrollment
* Active autoimmune disease (eg, rheumatoid arthritis, systemic lupus erythematosus, etc)
* Known pregnancy (no pregnancy testing will be performed)
* Overt acute illness/infection (according to Investigator's judgment) or febrile illness (temperature ≥ 38.0°C [100.4°F]) on the day of inclusion. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided for at least 2 consecutive days prior to enrollment
* Receipt of any vaccine within the 4 weeks preceding study enrollment
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Current or recent (within 3 weeks of enrollment) receipt of systemic antibiotics
* Use of chlorhexidine mouthwash for > 7 days within 3 weeks of enrollment
* Receipt of immunomodulators or immunosuppressive therapy, including long-term corticosteroid therapy
* Sub-gingival instrumentation/SRP within the 3 months prior to study enrollment

Note: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Serum titers of total anti-Porphyromonas gingivalis (Pg) antibody (Ab) | Day 01
Serum protease activity inhibition (PAI) titers | Day 01
Serum hemagglutination inhibition (HAI) titers | Day 01
Quantitative deoxyribonucleic acid (DNA)-based detection of Pg (saliva) | Day 01
DNA-based detection of Pg (sub-gingival plaque) | Day 01
Active-matrix metalloproteinase-8 (aMMP-8) levels measured by immunoassay in saliva (chairside assay) | Day 01

SECONDARY OUTCOMES:
Levels of inflammatory mediators (for example, cytokines, chemokines, matrix metalloproteinases) in serum measured by multiplex assay | Day 01
Levels of inflammatory mediators in saliva (including MMP-8) | Day 01
Salivary titers of total anti-Pg Ab | Day 01
Measurement of high sensitivity C-reactive protein (hsCRP) in serum | Day 01
Measurement of serum levels of pro-insulin | Day 01
Measurement of serum levels of c-peptide | Day 01
Measurement of serum levels of prostaglandin E2 (PGE2) | Day 01

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Iowa - Site Number : 8400002, Iowa City, Iowa
  - ADA Forsyth Institute Center for Clinical and Translational Research - Site Number : 8400004, Somerville, Massachusetts
  - Stony Brook School of Dental Medicine Periodontics Department- Site Number : 8400001, Stony Brook, New York
  - UT Health Houston School of Dentistry- Site Number : 8400003, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org